CLINICAL TRIAL: NCT06047366
Title: Buffered vs Unbuffered Local Anesthesia Using Lidocaine, Carbocaine, and Articaine in Mandibular Molars Diagnosed With Symptomatic Irreversible Pulpitis
Brief Title: Combination of Buffered Anesthetic to Treat Mandibular Molars
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Student PI is preparing for graduation and cannot complete the study as planned.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kenneth J. Spolnik DDS, Department of Endodontics Chair, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17799
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: lidocaine; articaine; mepivacaine; buffered local anesthetic; irreversible pulpitis
MeSH Terms: interventions — Sodium Bicarbonate; Epinephrine; Lidocaine; Carticaine; Mepivacaine

STUDY DESIGN:
Intervention Model Description: This study will be a single-center, controlled, randomized, double-blind (provider and subject), 2 treatment, 1 period, parallel study
Who Masked: Participant, Care Provider, Investigator
Masking Description: A statistician will provide a two-product randomization scheme which will randomize each of the 60 subjects on the order of their entry into the study. The research assistants will be aware of and document this scheme, but the student researcher/PI will not know what type of anesthetic will be administered.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buffered (Experimental): Buffered 2% lidocaine with 1:100,000 epinephrine Buffered 4% articaine with 1:100,000 epinephrine Buffered 3% mepivacaine Buffered local anesthetic (addition of sodium bicarbonate to make a 10% buffered solution)
  Interventions: Drug: Sodium bicarbonate; Drug: Lidocaine w/ epi; Drug: Articaine w/ epi; Drug: Mepivacaine plain
- Unbuffered (Active Comparator): Unbuffered 2% lidocaine with 1:100,000 epinephrine Unbuffered 4% articaine with 1:100,000 epinephrine Unbuffered 3% mepivacaine Standard local anesthetics
  Interventions: Drug: Lidocaine w/ epi; Drug: Articaine w/ epi; Drug: Mepivacaine plain

INTERVENTIONS:
Drug: Sodium bicarbonate — Onpharma's Onset sodium bicarbonate buffer to be added to a standard cartridge of dental local anesthetic
  Other Names: Onset Sodium Bicarbonate Inj., 8.4%, USP Neutralizing Additive Solutio
  Arms: Buffered
Drug: Lidocaine w/ epi — Septodont's standard formulation of 2% lidocaine with epinephrine
  Other Names: 2% lidocaine with 1:100,000 epinephrine
Drug: Articaine w/ epi — Septodont's standard formulation of 4% articaine with epinephrine
  Other Names: 4% articaine with 1:100,000 epinephrine
Drug: Mepivacaine plain — Septodont's standard formulation of 3% mepivacaine
  Other Names: 3% Mepivacaine

SUMMARY:
The purpose of this study is to determine whether a combination of anesthetics (numbing medicine) will adequately anesthetize teeth over a different combination. A second purpose is to see if the time needed to numb the nerve in a tooth is different between the two anesthetics.

DETAILED DESCRIPTION:
60 human subjects with Symptomatic Irreversible Pulpitis (SIP) in mandibular molars will be randomly allocated into 2 groups. One group will receive a combination of: 1 cartridge of buffered 2% lidocaine w/ 1:100k epi via inferior alveolar nerve block (IANB) followed by 1 cartridge of 3% mepivacaine via IANB. This will be followed by 0.5 cartridges (0.9mL) of buffered 4% articaine with 1:100k epi via buccal infiltration and 0.5 cartridges of buffered 4% articaine with 1:100k epi via lingual infiltration. All IANB injections will include a lingual block. The second group will be provided an unbuffered version of the same combination. An electronic pulp tester (EPT) will be used to determine the vitality of the treated tooth. Endodontic treatment will be initiated after two consecutive EPT readings of 80, displaying pulpal anesthesia. Profound pulpal anesthesia is described by the patient's report on the visual analog scale after the pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 80 years old
* Have the ability and willingness to independently consent to treatment and study participation
* Have an uncomplicated medical history (ASA I and II)
* Not be pregnant
* Have no allergies local anesthetics/sulfites (confirmed or self-reported)
* Not be taking any medications that may affect the proper assessment of the anesthetic (no acetaminophen or short-acting NSAIDs such as ibuprofen within the previous 6 hours; no long-acting NSAIDs such as naproxen within the previous 16 hours)
* Not require nitrous oxide during treatment, and the injection area should appear healthy with no other pre-existing conditions or infections that may compromise an accurate collection of data
* Be experiencing signs of irreversible pulpitis (an exaggerated response to cold that lingers longer than 10 seconds) in a mandibular molar at the time of conducting the study

Exclusion Criteria:

* A negative response to cold in the proposed treatment tooth
* A radiographic periradicular pathosis more advanced than a widened periodontal ligament or have an intraoral swelling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Spolnik, DDS, Study Chair — Program Director
Locations (1):
- ndiana University School of Dentistry Graduate Endodontics Dept., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg PA, Amin KG, Zibari Y, Lin LM. Comparison of 4% articaine with 1:100,000 epinephrine and 2% lidocaine with 1:100,000 epinephrine when used as a supplemental anesthetic. J Endod. 2007 Apr;33(4):403-5. doi: 10.1016/j.joen.2006.11.019. Epub 2007 Feb 20. PMID 17368327
- [Background] Goodis HE, Poon A, Hargreaves KM. Tissue pH and temperature regulate pulpal nociceptors. J Dent Res. 2006 Nov;85(11):1046-9. doi: 10.1177/154405910608501114. PMID 17062748
- [Background] Christoph RA, Buchanan L, Begalla K, Schwartz S. Pain reduction in local anesthetic administration through pH buffering. Ann Emerg Med. 1988 Feb;17(2):117-20. doi: 10.1016/s0196-0644(88)80293-2. PMID 2827545
- [Background] Schellenberg J, Drum M, Reader A, Nusstein J, Fowler S, Beck M. Effect of Buffered 4% Lidocaine on the Success of the Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Randomized, Double-blind Study. J Endod. 2015 Jun;41(6):791-6. doi: 10.1016/j.joen.2015.02.022. Epub 2015 Apr 1. PMID 25841959
- [Background] Saatchi M, Farhad AR, Shenasa N, Haghighi SK. Effect of Sodium Bicarbonate Buccal Infiltration on the Success of Inferior Alveolar Nerve Block in Mandibular First Molars with Symptomatic Irreversible Pulpitis: A Prospective, Randomized Double-blind Study. J Endod. 2016 Oct;42(10):1458-61. doi: 10.1016/j.joen.2016.07.004. Epub 2016 Aug 6. PMID 27507627
- [Background] Fowler S, Reader A. Is a volume of 3.6 mL better than 1.8 mL for inferior alveolar nerve blocks in patients with symptomatic irreversible pulpitis? J Endod. 2013 Aug;39(8):970-2. doi: 10.1016/j.joen.2013.04.007. Epub 2013 May 16. PMID 23880260
- [Background] Kanaa MD, Whitworth JM, Meechan JG. A prospective randomized trial of different supplementary local anesthetic techniques after failure of inferior alveolar nerve block in patients with irreversible pulpitis in mandibular teeth. J Endod. 2012 Apr;38(4):421-5. doi: 10.1016/j.joen.2011.12.006. Epub 2012 Feb 2. PMID 22414822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buffered | Unbuffered
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buffered | Unbuffered | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [28 to 47] | 28 [23 to 49] | 33.5 [23 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Median Visual Analogue Scale (VAS) Score as a Measure of Profoundness of Pulpal Anesthesia
Description: Patient will report their comfort during treatment based on a visual analogue scale (VAS) graphic. Visual analog scale (VAS) is based on a scale of 0-10 related to patient comfort. A VAS score of 10 would mean the patient was extremely uncomfortable during treatment indicating there was inadequate anesthesia. A VAS score of 0 indicates no pain.
Time Frame: Up to 20 minutes post-drug administration
Population: Patients who achieved profound pulpal anesthesia
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Buffered | Unbuffered
Number analyzed (Participants) | 17 | 15
units on a scale | 0 [0 to 2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Buffered vs Unbuffered; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney) — p < 0.05 was used as the threshold for statistical significance

2. Secondary Outcome: Median Time to Profound Pulpal Anesthesia
Description: An electronic pulp tester will be used to assess anesthesia after anesthetic is administered. The median time needed to achieve profound pulpal anesthesia for the two groups will be calculated using the Kaplan-Meier method and compared with a log-rank test, with patients who failed to achieve profound pulpal anesthesia censored at 15 minutes.
Time Frame: Up to 15 minutes post-drug administration
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Buffered | Unbuffered
Number analyzed (Participants) | 20 | 20
minutes | 5.28 [4.22 to 6.17] | 7.96 [5.50 to 10.15]
Statistical Analysis 1: Comparison: Buffered vs Unbuffered; Test type: Other; p = 0.09, Log Rank — p < 0.05 was used as the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: during a single visit, up to two hours
Arm/Group | Buffered | Unbuffered
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT06047366/Prot_SAP_000.pdf